CLINICAL TRIAL: NCT04213365
Title: Management of Cognitive Difficulties After Cancer Treatments in Women Treated for Breast Cancer: Feasibility Study (Step 1 of the Cog-Stim Protocol)
Acronym: COG STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A02500-57
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cognitive stimulation and adapted physical activity (Other): 12 weeks of cognitive stimulation sessions coupled with APA (Adapted Physical Activity) sessions.
  Interventions: Other: Cognitive stimulation sessions coupled with Adapted Physical Activity sessions.

INTERVENTIONS:
Other: Cognitive stimulation sessions coupled with Adapted Physical Activity sessions. — 12 weeks of cognitive stimulation sessions coupled with APA (Adapted Physical Activity) sessions.

SUMMARY:
Investigator general objective is therefore to study and compare the benefit of several methods of management of cognitive difficulties reported by patients during treatment for breast cancer, among several treatments, offered independently in patients' homes and supervised from a distance: adapted physical activity only, cognitive stimulation only, and adapted physical activity coupled with cognitive stimulation (during separate sessions). The study will therefore be the first to include a group benefiting from these two management methods, which will make it possible to assess the individual benefit of cognitive stimulation sessions and adapted physical activity but also the benefit of combined sessions.As this type of combined management has never been the subject of a study, and previous studies relating to a single type of management having raised patient adhesion difficulties, it does not seem certain that this type of care is feasible in practice. Before studying its effectiveness, it is therefore essential to check the feasibility and acceptability of such a program combining sessions of adapted physical activity and cognitive stimulation sessions.Investigator will therefore first carry out a feasibility study, longitudinal and monocentric, which will assess the adherence of patients treated for breast cancer to the performance of cognitive stimulation sessions coupled with sessions of adapted physical activity.This feasibility study is a key stage of the Cog-Stim protocol because its results will probably highlight the obstacles to the intervention program, which will allow the investigator to propose adjustments to improve the study design for the following stages of the protocol. (design optimization).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18,
* Patient with localized breast cancer, starting or receiving adjuvant radiotherapy , having or not receiving previous adjuvant chemotherapy, not yet having started hormone therapy,
* Patient with a cognitive complaint having a significant impact on her quality of life (FACT
* Cog questionnaire, QoL score ≤ percentile 10 by age),
* Absence of major cognitive impairment preventing the performance of cognitive tests (compliance with the MoCA score threshold according to the age and educational level of the patient according to GRECOGVASC standards)
* Absence of personality disorders and known progressive psychiatric pathology (e.g. schizophrenia),
* Absence of symptomatic neurological history (neurological sequelae of a head trauma, stroke with loss of consciousness> 30 min, multiple sclerosis, epilepsy, neurodegenerative pathology, etc.),
* Patient with level of education 3 "end of primary education" minimum (Barbizet scale),
* Have access to a computer (fixed or portable) equipped with a keyboard, a webcam (or the possibility of connecting one), headphones or speakers; have an internet connection and an e-mail account; be able to use these tools and Equipment,
* Mastery of the French language,
* Patient who signed the consent to participate in the study.
* Patients should start the study during radiation therapy.

Exclusion Criteria:

* Abuse of alcohol or drug use,
* Severe visual and / or hearing loss,
* Patient unable to respond to cognitive tests,
* Medical contraindication to the practice of adapted physical activity
* Cognitive management in progress,
* Patient's refusal to participate,
* Patient deprived of liberty or under guardianship,
* Patient unable to submit to study monitoring for geographic, social or psychopathological reasons.

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Patient adherence | between inclusion and 3 months
  The proposrtion of patients who will realize cognitive stimulation sessions coupled with sessions of adapted physical activity

SECONDARY OUTCOMES:
Proportion of acceptance | Before inclusion
  Proportion of patient who accept the participation in the study
Patient satisfaction | between inclusion and 3 months
  Satisfaction questionnary (Patient satisfaction questionnary; minimum 1 t maximum 5; 15 questions)

CONTACTS AND LOCATIONS:
Locations (1):
- centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Binarelli G, Joly F, Christy F, Clarisse B, Lange M. Digital multimodal intervention for cancer-related cognitive impairment in breast-cancer patients: Cog-Stim feasibility study. BMC Psychiatry. 2025 Mar 17;25(1):249. doi: 10.1186/s12888-025-06630-9. PMID 40098149